CLINICAL TRIAL: NCT06042517
Title: Mechanisms of Ultrasound Neuromodulation Effects in Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000034954; 1R01DK131127-01A1 (NIH)
Record Dates: First submitted 2023-08-22; First posted 2023-09-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Ultrasonography; Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: For Cohort 4: T2DM subjects, age-, BMI- and HbA1c-matched to cohorts 1 and 2 will be recruited from the same pool of volunteers and selected according to the same inclusion and exclusion criteria outlined in the human subject protection plan.
  5 additional subjects will be recruited to participate in cohort 3.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Cohort 1: Ultrasound during a hyperinsulinemic euglycemic clamp (HEC). (Experimental): Hepatic ultrasound during a hyperinsulinemic euglycemic clamp (HEC).
  Interventions: Device: Ultrasound; Diagnostic Test: CGM glucose reading; Diagnostic Test: HEC - Hyperinsulinemic-Euglycemic-Clamp
- Cohort 2: Ultrasound then NMR with unlabeled glucose. (Experimental): Hepatic ultrasound and subsequent NMR measurement of glycogen with unlabeled glucose.
  Interventions: Device: Ultrasound; Diagnostic Test: OGTT with unlabeled glucose and liver NMR; Diagnostic Test: CGM glucose reading
- Cohort 3: Ultrasound then NMR with carbon13 labeled glucose. (Experimental): Hepatic ultrasound and subsequent NMR measurement of glycogen with carbon13 labeled glucose.
  Interventions: Device: Ultrasound; Diagnostic Test: OGTT with carbon-13 labeled glucose and liver NMR; Diagnostic Test: CGM glucose reading
- Cohort 4: Dual site ultrasound stimulation followed by CGM glucose recording alone. (Experimental): Hepatoportal plexus + superior mesenteric plexus dual site ultrasound stimulation followed by CGM glucose recording alone.
  Interventions: Device: Ultrasound; Diagnostic Test: CGM glucose reading

INTERVENTIONS:
Device: Ultrasound — The General Electric LOGIQ E10 ultrasound pulsed doppler imaging system and C1-6-D XDclear abdominal curvilinear probe will be used to administer ultrasound.
Diagnostic Test: OGTT with unlabeled glucose and liver NMR — Subjects will undergo an OGTT with unlabeled glucose to measure liver glycogen concentration by NMR spectroscopy.
  Arms: Cohort 2: Ultrasound then NMR with unlabeled glucose.
Diagnostic Test: OGTT with carbon-13 labeled glucose and liver NMR — Subjects will undergo an OGTT with carbon-13 labeled glucose to measure liver glycogen synthesis rate by NMR spectroscopy.
  Arms: Cohort 3: Ultrasound then NMR with carbon13 labeled glucose.
Diagnostic Test: CGM glucose reading — A continuous glucose monitor (CGM) will be collecting glucose level changes over a 10-14day time period after the ultrasound.
Diagnostic Test: HEC - Hyperinsulinemic-Euglycemic-Clamp — A constant i.v. insulin and variable glucose infusion will be used to determine insulin sensitivity of study participants.
  Arms: Cohort 1: Ultrasound during a hyperinsulinemic euglycemic clamp (HEC).

SUMMARY:
This study aims to evaluate the effect of hepatic ultrasound treatment on changes from baseline in whole-body insulin sensitivity during a hyperinsulinemic, euglycemic clamp (HE Clamp).

DETAILED DESCRIPTION:
Drop-outs will be replaced; data will be used as much as can be. Subjects will undergo a Screening visit to assess eligibility and will then be scheduled to undergo 2 outpatient US treatment visits.

On day three subjects first undergo a third ultrasound session and then will either undergo Oral Glucose Tolerance Test (OGTT) with carbon13 (13C-glucose) tracer administration and subsequent NMR spectroscopy OR if enrolled into the HEC study arm will undergo euglycemic clamp testing. Following these procedures there will be an approximately two-week follow-up observational Period (with CGM). A two-week washout period will be followed by another cycle of the same procedures of either OGTT/NMR or HEC study, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic (T2D) subjects must be aged 18-80 and must be able to provide written informed consent
* All subjects must have had T2D for at least 3 months prior to study enrollment. All subjects must be either on diet and exercise or oral antidiabetic agents alone, not on insulin or any form of insulin or GLP-1 receptor agonists.
* Subjects must demonstrate:

  1. A past medical history of abnormal glucose control and carry a diagnosis of T2D according to current ADA criteria:

     * A fasting plasma glucose (FPG) level of 126 mg/dL (7.0 mmol/L) or higher, or
     * A 2-hour plasma glucose level of 200 mg/dL (11.1 mmol/L) or higher during a 75-g oral glucose tolerance test (OGTT), or
     * A random plasma glucose of 200 mg/dL (11.1 mmol/L) or higher in a patient with classic symptoms of hyperglycemia or hyperglycemic crisis or
     * A hemoglobin A1c (HbA1c) level of 6.5% or higher.
  2. Be willing to carry a continuous glucose monitor for at least 10 days.
  3. Be willing to follow all required instructions by study personnel and appear for the required laboratory assessments, including euglycemic clamps and OGTT.

Exclusion Criteria:

* BMI >40kg/m2.
* Untreated proliferative retinopathy
* Creatinine clearance < 60 ml/min/1.73 m2.
* Serum creatinine ≥1.5 mg/dL
* Positive pregnancy test, or presently breast-feeding, or failure to follow effective contraceptive measures
* Active infection including hepatitis C, hepatitis B, HIV,
* Any history of Active alcohol abuse
* History of non-adherence to prescribed regimens
* Baseline Hgb < 10.5 g/dL in females, or < 13 g/dL in males
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy (low-dose aspirin treatment is allowed)
* Co-existing cardiac disease with active medication titration. Patients on stable meds without active cardiac complications permitted.
* Liver function tests outside of 3xUL of normal range
* GI disorders potentially interfering with the ability to absorb oral medications and h/o upper GI surgery that might have changed anatomy in the target areas.
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | Measured during HE clamp.
  Insulin Sensitivity calculated as Glucose disposal rate / insulin ratio during steady state (M/I) to evaluate the effect of hepatic ultrasound treatment on changes from baseline in whole-body insulin sensitivity during a hyperinsulinemic, euglycemic clamp (HE Clamp)
Glucose disposal rate | Measured during HE clamp.
  Glucose disposal rate during steady state (M) to evaluate the effect of hepatic ultrasound treatment on changes from baseline in whole-body insulin sensitivity during a hyperinsulinemic, euglycemic clamp (HE Clamp)
Glucose metabolic clearance rate | Measured during HE clamp.
  Glucose metabolic clearance rate during steady state (MCR) to evaluate the effect of hepatic ultrasound treatment on changes from baseline in whole-body insulin sensitivity during a hyperinsulinemic, euglycemic clamp (HE Clamp)

SECONDARY OUTCOMES:
Absolute glycogen level | during glucose tolerance testing (for 180 minutes).
  The effect of hepatic plexus-directed pFUS on absolute glycogen level by observing the metabolic fate of unlabeled glucose ingested during oral glucose tolerance testing measured by 13C liver NMR-spectroscopy.
Glycogen synthesis rates | during glucose tolerance testing (for 180 minutes).
  Glycogen synthesis rates are derived from plasma 13C -glucose levels achieved during the OGTT and subsequent appearance of 13C -tracer in liver glycogen
Change from baseline in blood glucose (BG) time spent in defined glucose ranges | 1 week
  Change from baseline in blood glucose (BG) time spent in defined glucose ranges assessed using a continuous glucose monitoring system (CGMS)
Average daily glucose | 1 week
  Average daily glucose assessed using a continuous glucose monitoring system (CGMS)
Low blood glucose index (LBGI) | 1 week
  Frequency of low glucose events detected during continuous glucose measurement.
High blood glucose index (HBGI) | 1 week
  Frequency of high glucose events detected during continuous glucose measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No